CLINICAL TRIAL: NCT04833881
Title: Proteomics/Modifier Based on Mass Spectrometry Reveals the Pathogenesis of Eclampsia During Pregnancy and the Screening of Disease Markers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xiaoke Wu, Professor and Director of Obstetrics and Gynecology Department, Heilongjiang University of Chinese Medicine
Other Study IDs: PREECLAMPSIA
Record Dates: First submitted 2021-03-11; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Mechanism; Marker Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The control group
- Experimental group

INTERVENTIONS:
Other:

SUMMARY:
Pregnancy-induced hypertension is a unique abnormal blood pressure disease in women during pregnancy, including eclampsia, preeclampsia, pregnancy-induced hypertension, chronic hypertension and so on. Eclampsia can lead to convulsions, proteinuria, multiple organ failure, and eventually death. It is a very serious disease in women, and the incidence of pregnancy-induced hypertension during pregnancy is between 4% and 10%. The incidence of eclampsia ranges from 2% to 5%. Studies have shown that there are about 60,000 cases of stillbirth or stillbirth due to eclampsia every year worldwide. At present, there are many theories about the pathogenesis of eclampsia, such as oxidative stress theory, maternal and fetal interaction theory, immune imbalance theory, heredity theory and so on.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women with preeclampsia:

  1. Singleton women who meet the diagnostic criteria for preeclampsia.
  2. No previous history of major disease.
  3. Body mass index is between 23-25kg/m2.
  4. 20-45 years old.
  5. 22-42 weeks of gestation.
  6. Participate in the test voluntarily and sign the informed consent.

  2. Healthy pregnant women:
  1. In good health, no history of major diseases before pregnancy, pregnant women and single mothers with healthy fetuses (newborn) after pregnancy and delivery.
  2. Body mass index is between 23-25kg/m2.
  3. 20-45 years old.
  4. 22-42 weeks of gestation.
  5. Participate in the test voluntarily and sign the informed consent.

     Exclusion Criteria:
* 1. Women with preeclampsia:

  1. Patients with essential hypertension.
  2. Pregnant women with high blood glucose before and/or during pregnancy.
  3. Convulsions on the basis of preeclampsia that cannot be explained by other reasons.
  4. Women with primary disease due to other non-preeclampsia diseases before and after pregnancy, such as cardiovascular, cerebrovascular, liver, kidney, hematopoietic, endocrine, immune, precancerous lesions or cancers, including the reproductive system.
  5. Twin or multiple births.
  6. Pregnant women with mental disorders or mental diseases.
  7. Using illegal drugs before and after pregnancy.
  8. Persons with sexually transmitted diseases or infectious diseases.
  9. Pregnant women receiving prenatal steroid therapy.

  2. Healthy pregnant women:
  1. Patients with severe maternal and/or fetal (newborn) adverse events during or after the third trimester of pregnancy or delivery. Such as intrauterine infection, amniotic fluid embolism and other serious maternal adverse events; Fetal malformation, fetal growth restriction, fetal intrauterine distress, neonatal hemolysis and other serious fetal (neonatal) adverse events.
  2. Pregnant women with other diseases before and after pregnancy, such as cardiovascular and cerebrovascular, liver, kidney, hematopoietic system, endocrine system, immune system, precancerous lesions or cancer, including the reproductive system, and other serious primary diseases.
  3. Women with a clear cause of premature delivery.
  4. Twin or multiple births.
  5. Pregnant women with mental disorders or mental diseases.
  6. Use illegal drugs before and after pregnancy.
  7. Persons suffering from sexually transmitted diseases or infectious diseases.
  8. Pregnant women receiving prenatal steroid therapy.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Women with preeclampsia:
  1. Singleton women who meet the diagnostic criteria for preeclampsia.
  2. No previous history of major disease.
  3. Body mass index is between 23-25kg/m2.
  4. 20-45 years old.
  5. 22-42 weeks of gestation.
  6. Participate in the test voluntarily and sign the informed consent.
  2. Healthy pregnant women:
  1. In good health, no history of major diseases before pregnancy, pregnant women and single mothers with healthy fetuses (newborn) after pregnancy and delivery.
  2. Body mass index is between 23-25kg/m2.
  3. 20-45 years old.
  4. 22-42 weeks of gestation.
  5. Participate in the test voluntarily and sign the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Proteomics and acetylation modification analysis of placenta, blood, urine, and cervical secretions | 2023-08
  Proteomics analysis is carried out using the TMT labeling quantitative method, the significantly differentially expressed proteins and modification sites are screened out, and then the proteins with significantly different changes are used as disease signs; Through the GO classification analysis of the protein, the subcellular structure location analysis of the protein is carried out, and the mitochondrial-related protein and skeleton protein are concerned. Through the enrichment of acetylated antibody modified protein-peptide, the changes of modified protein and its regulatory mechanism were analyzed, and the regulatory role of acetylated protein in mitochondrial metabolism and immune response was found. This study uses the Mfuzz clustering method to perform clustering analysis of the expression profile of proteins, the pathogenesis of the disease through protein enrichment analysis, pathway analysis, and interaction analysis are explored.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: Undecided